CLINICAL TRIAL: NCT06517602
Title: Effect of Daily Consumption of Moringa Oleifera Leaves on Glycemic Control of Saharawi Women With Type 2 Diabetes
Brief Title: Effect of Moringa Oleifera Leaves on Glycemic Control of Women With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Alberto Battezzati, Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-11-2018
Record Dates: First submitted 2024-07-11; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes
Keywords: Moringa oleifera; Type 2 diabetes; Humans; Glucose; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moringa (Experimental): The experimental group received for 3 months a daily supplementation of 10g of Moringa oleifera leaf powder to consume within the two main meals.
  Interventions: Dietary Supplement: Supplementation of Moringa oleifera leaf powder
- Control (No Intervention): The control group were asked to refrain from consuming Moringa oleifera leaves throughout the study period (3 months).

INTERVENTIONS:
Dietary Supplement: Supplementation of Moringa oleifera leaf powder — Women in the experimental group were asked to consistently take the prescribed oral hypoglycemic therapy and to maintain their lifestyle and eating habits. In addition, for the duration of the study (3 months), the experimental group was provided with 10 g of Moringa oleifera leaf powder daily to be consumed with main meals.
  Arms: Moringa

SUMMARY:
The objective of this clinical trial was to understand whether supplementation of Moringa oleifera leaf powder improved glycemic management in Sahrawi women with type 2 diabetes living in refugee camps. The main question sought to be answered was:

- Does daily supplementation of Moringa oleifera leaf powder, in addition to oral hypoglycemic therapy, improve glycosylated hemoglobin and fasting blood glucose?

Researchers compared Moringa supplementation with no Moringa consumption to see if Moringa oleifera worked to improve glycemic control.

Participants had to:

* Take Moringa oleifera leaves daily or abstain from consuming Moringa for 3 months.
* Consistently take prescribed oral hypoglycemic agents
* Undergo clinical examinations and measurement of biochemical, metabolic and body composition parameters at the time of recruitment and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes for at least 1 year
* Absence of advanced retinopathy, terminal renal failure, active diabetic ulcers, amputations, and heart failure
* Treatment with only oral hypoglycemic drugs.

Exclusion Criteria:

* Diagnosis of type 1 diabetes
* Pregnancy or lactation
* Treatment with insulin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-02-23 (Actual); Study Completion 2020-02-23 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | Glycosylated hemoglobin was measured at recruitment and at the end of the study (three months)
Fasting glucose | Fasting glucose was measured at recruitment and at the end of the study (three months)

SECONDARY OUTCOMES:
BMI | BMI were measured at recruitment and at the end of the study (3 months)
Waist circumference | Waist circumference were measured at recruitment and at the end of the study (3 months)
Hip circumference | Hip circumference were measured at recruitment and at the end of the study (3 months)
% body fat | % of body fat were measured at recruitment and at the end of the study (3 months)
Blood pressure | Systolic and diastolic blood pressure were measured at recruitment and at the end of the study (3 months)
  Systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Dispensaris of Edchedería, Bir Lehlu, Mahbes, and Farsia (Smara camp), Tindouf, Algeria